CLINICAL TRIAL: NCT02871908
Title: Lactobacillus Reuteri DSM 17938 in the Prevention of Antibiotic-associated Diarrhea in Children: Protocol of a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Hanna Szajewska, Professor and Chair of Pediatrics at the Medical University of Warsaw, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12/08/2016
Record Dates: First submitted 2016-08-16; First posted 2016-08-18 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Diarrhea; Antibiotic Associated Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L reuteri DSM 17938 (Experimental): L reuteri DSM 17938 2 x 10^8 twice daily
  Interventions: Drug: Lactobacillus reuteri DSM 17938
- Controls (Placebo Comparator): Identically appearing placebo twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus reuteri DSM 17938 — Lactobacillus reuteri DSM 17938 twice daily 2 x 10^8
  Arms: L reuteri DSM 17938
Drug: Placebo — Placebo
  Arms: Controls

SUMMARY:
The aim of this study is to assess the effect of Lactobacillus reuteri DSM 17938 administration for the prevention of diarrhea and AAD in children.

DETAILED DESCRIPTION:
Introduction:

Addition of some probiotics appears to reduce the risk of antibiotic-associated diarrhea (AAD). Effects of probiotics are strain specific, thus the efficacy and safety of each probiotic strain should be established separately. We aim to assess the effect of Lactobacillus reuteri DSM 17938 administration for the prevention of diarrhea and AAD in children.

Methods and analysis:

A total of 250 children younger than 18 years treated with antibiotics will be enrolled into a double-blind, randomized placebo-controlled trial in which they will additionally receive L reuteri DSM 17938 at a dose 2 x 10^8 colony-forming units or an identically appearing placebo, orally, twice daily, for the entire duration of antibiotic treatment. The primary outcome measures will be the frequency of diarrhea and AAD. Diarrhea will be defined according to one of 3 definitions: (a) ≥3 loose or watery stools per day for a minimum of 48 hours during antibiotic treatment; (b) ≥3 loose or watery stools per day for a minimum of 24 hours during antibiotic treatment; (c) ≥2 loose or watery stools per day for a minimum of 24 hours during antibiotic treatment. AAD will be diagnosed in cases of diarrhea, defined clinically as above, caused by C. difficile or for otherwise unexplained diarrhea (i.e. negative laboratory stool tests for infectious agents).

ELIGIBILITY:
Inclusion Criteria:

* age younger than 18 years;
* oral or intravenous antibiotic therapy which started within 24 hours of enrollment;
* signed informed consent.

Exclusion Criteria:

* pre-existing acute or chronic diarrhea,
* history of chronic gastrointestinal disease (e.g., inflammatory bowel disease, cystic fibrosis, celiac disease, food allergy) or other severe chronic disease (e.g., neoplastic diseases), immunodeficiency,
* use of probiotics within 2 weeks prior to enrollment,
* use of antibiotics within 4 weeks prior to enrollment,
* prematurity, and exclusive breastfeeding.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
frequencies of diarrhea and antibiotic associated diarrhea | during antibiotic treatment, an average of 10 days and 7 days of follow up
  Three different definitions of diarrhea will be used, as the definitions of diarrhea/AAD in published studies vary. These will include diarrhea defined as: (a) ≥3 loose or watery stools per day for a minimum of 48 hours during antibiotic treatment; (b) ≥3 loose or watery stools per day for a minimum of 24 hours during antibiotic treatment, and (c) ≥2 loose or watery stools per day for a minimum of 24 hours during antibiotic treatment. AAD will be diagnosed in cases of diarrhea, defined clinically as above, caused by C. difficile or for otherwise unexplained diarrhea (i.e., negative laboratory stool tests for infectious agents). In all cases, loose or watery stools will correspond to scores of 5 to 7 on the BSF scale or A-consistency on the AISS.

SECONDARY OUTCOMES:
infectious diarrhea | during antibiotic treatment, an average of 10 days and 7 days of follow up
  rotavirus, adenovirus, norovirus, Salmonella, Shigella, Campylobacter, Yersinia and C. difficile
the need for discontinuation of the antibiotic treatment | during antibiotic treatment, an average of 10 days
the need for hospitalization to manage the diarrhea (in outpatients) | during antibiotic treatment, an average of 10 days and 7 days of follow up
the need for intravenous rehydration in any of the study groups | during antibiotic treatment, an average of 10 days and 7 days of follow up
adverse events | during antibiotic treatment, an average of 10 days and 7 days of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatrics, The Medical University of Warsaw, Poland, Warsaw, Poland

REFERENCES:
- [Derived] Kolodziej M, Szajewska H. Lactobacillus reuteri DSM 17938 in the prevention of antibiotic-associated diarrhoea in children: protocol of a randomised controlled trial. BMJ Open. 2017 Jan 5;7(1):e013928. doi: 10.1136/bmjopen-2016-013928. PMID 28057659